CLINICAL TRIAL: NCT01778010
Title: Modafinil in a Human Laboratory Model of Cocaine Relapse
Brief Title: Modafinil for Smoked Cocaine Self-Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5738; R01DA023650 (NIH)
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Cocaine Dependence
Keywords: cocaine; modafinil; self-administration; DRD4
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil; Cocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Modafinil 0mg + Cocaine 0, 12, 25, 50 mg (Placebo Comparator): Participants were maintained on modafinil (0 mg/day) for 15 days, and underwent a dose response of cocaine.
  Interventions: Drug: Modafinil 0 mg; Drug: Cocaine 0 mg; Drug: Cocaine 12 mg; Drug: Cocaine 25 mg; Drug: Cocaine 50 mg
- Modafinil 200mg + Cocaine 0, 12, 25, 50 mg (Experimental): Participants were maintained on modafinil (200 mg/day) for 15 days, and underwent a dose response of cocaine.
  Interventions: Drug: Modafinil 200 mg; Drug: Cocaine 0 mg; Drug: Cocaine 12 mg; Drug: Cocaine 25 mg; Drug: Cocaine 50 mg
- Modafinil 400mg + Cocaine 0, 12, 25, 50 mg (Experimental): Participants were maintained on modafinil (400 mg/day) for 15 days, and underwent a dose response of cocaine.
  Interventions: Drug: Modafinil 400 mg; Drug: Cocaine 0 mg; Drug: Cocaine 12 mg; Drug: Cocaine 25 mg; Drug: Cocaine 50 mg

INTERVENTIONS:
Drug: Modafinil 0 mg — Modafinil (0 mg/day)
  Arms: Modafinil 0mg + Cocaine 0, 12, 25, 50 mg
Drug: Modafinil 200 mg — Modafinil (200 mg/day)
  Arms: Modafinil 200mg + Cocaine 0, 12, 25, 50 mg
Drug: Modafinil 400 mg — Modafinil (400 mg/day)
  Arms: Modafinil 400mg + Cocaine 0, 12, 25, 50 mg
Drug: Cocaine 0 mg — Cocaine (0 mg/day)
Drug: Cocaine 12 mg — Cocaine (12 mg/day)
Drug: Cocaine 25 mg — Cocaine (25 mg/day)
Drug: Cocaine 50 mg — Cocaine (50 mg/day)

SUMMARY:
Modafinil has been reported to reduce cocaine use in a clinical sample of infrequent users (2 days/week), but the effects of modafinil on cocaine self-administration in the laboratory have not been studied. The present study investigated the effects of modafinil maintenance on cocaine self-administration by frequent users (4 days/week) under controlled laboratory conditions. During this 48-day double-blind, crossover design study, the effects of modafinil maintenance (0, 200, and 400mg/day) on response to smoked cocaine (0, 12, 25, and 50 mg) were examined in nontreatment seeking cocaine-dependent individuals (n = 8).

ELIGIBILITY:
Inclusion Criteria:

1. Smokes cocaine
2. Has patterns of smoked cocaine use in terms of frequency and amount which parallel or exceed those administered in the study.
3. Age 21-50.
4. Able to give informed consent, and comply with study procedures.
5. Normal body weight Within normal weight range (for appropriate frame) according to 1983 Metropolitan Weight tables -

Exclusion Criteria:

1. Current seizure disorder, heart disease or a history of serious adverse effects due to cocaine.
2. Dependence on substances (other than cocaine or nicotine) or a history of dependence on alcohol
3. Request for drug treatment
4. Judged to be noncompliant with study protocol.
5. Current use of any psychotropic medication.
6. Clinical laboratory tests outside normal limits that are clinically unacceptable to the study physician (BP > 140/90; BUN, creatinine, LFTs > 3x ULN; hematocrit < 34 for women, < 36 for men; pseudocholinesterase deficiency)
7. History of myocardial infarction or ischemia, clinically significant left ventricular hypertrophy, angina, clinically significant arrhythmia, or mitral valve prolapse
8. Currently meeting DSM-IV criteria for all major psychiatric/psychotic disorders other than transient psychosis due to drug abuse
9. Current parole or probation Self-report during interview -

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — NYS Psychiatric Institute
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Modafinil + Cocaine: During this within-subjects, alternating in-patient/outpatient 48-day study, participants were maintained on modafinil (placebo, 200, and 400mg/day) and underwent a dose response of smoked cocaine (0, 12, 25, and 50mg).
Period: Overall Study
Arm/Group | Modafinil + Cocaine
Started | 13
Completed | 8
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — abnormal ECG before meds | 1
Not completed — Arrested | 1
Not completed — rash while on placebo | 1

BASELINE CHARACTERISTICS:
Population: During this within-subjects, alternating in-patient/outpatient 48-day study, participants were maintained on modafinil (placebo, 200, and 400mg/day) and four doses of smoked cocaine (0, 12, 25, and 50mg).
Groups:
- Modafinil + Cocaine: During this within-subjects, alternating in-patient/outpatient 48-day study, participants were maintained on modafinil (placebo, 200, and 400mg/day) and four doses of smoked cocaine (0, 12, 25, and 50mg).
Arm/Group | Modafinil + Cocaine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Self-administration
Description: The number of purchased cocaine doses as a function of cocaine dose and modafinil maintenance condition.
Time Frame: 48 days
Population: Eight patients contributed to each condition, in a within-subjects manner.
Measure: Mean (Standard Error); unit: Number of doses purchased
Groups:
- Modafinil 0mg + Cocaine 0mg; Modafinil 200mg + Cocaine 0mg; Modafinil 400mg + Cocaine 0mg; Modafinil 0mg + Cocaine 12mg; Modafinil 200mg + Cocaine 12mg; Modafinil 400mg + Cocaine 12mg; Modafinil 0mg + Cocaine 25mg; Modafinil 200mg + Cocaine 25mg; Modafinil 400mg + Cocaine 25mg; Modafinil 0mg + Cocaine 50mg; Modafinil 200mg + Cocaine 50mg; Modafinil 400mg + Cocaine 50mg: During this within-subjects, alternating in-patient/outpatient 48-day study, participants were maintained on modafinil (placebo, 200, and 400mg/day) and four doses of smoked cocaine (0, 12, 25, and 50mg).
Arm/Group | Modafinil 0mg + Cocaine 0mg | Modafinil 200mg + Cocaine 0mg | Modafinil 400mg + Cocaine 0mg | Modafinil 0mg + Cocaine 12mg | Modafinil 200mg + Cocaine 12mg | Modafinil 400mg + Cocaine 12mg | Modafinil 0mg + Cocaine 25mg | Modafinil 200mg + Cocaine 25mg | Modafinil 400mg + Cocaine 25mg | Modafinil 0mg + Cocaine 50mg | Modafinil 200mg + Cocaine 50mg | Modafinil 400mg + Cocaine 50mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Number of doses purchased | 0 (0) | 0 (0) | 0 (0) | 2.2 (0.3) | 1.5 (0.3) | 2.1 (0.1) | 4.1 (0.2) | 2.5 (0.3) | 2.6 (0.3) | 4.5 (0.1) | 3.5 (0.3) | 3 (0.3)

2. Secondary Outcome: Drug Quality Cluster
Description: Visual analogue scale ratings on the 'Drug Quality' cluster as a function of cocaine dose and modafinil maintenance condition. A cluster score was derived by taking the arithmetic average of the items in the cluster. Scores range from 0-100, with higher scores indicating greater agreement with the term. The "Drug Quality Cluster" consisted of three items:
  1. "the choice was of high quality"
  2. "the choice was potent"
  3. "I liked the choice" Higher scores indicate increasing agreement with the statement, which would indicate a poorer outcome.
Time Frame: 48 days
Population: Eight subjects participants in each condition in a within-subjects fashion.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Modafinil 0mg + Cocaine 0mg | Modafinil 200mg + Cocaine 0mg | Modafinil 400mg + Cocaine 0mg | Modafinil 0mg + Cocaine 12mg | Modafinil 200mg + Cocaine 12mg | Modafinil 400mg + Cocaine 12mg | Modafinil 0mg + Cocaine 25mg | Modafinil 200mg + Cocaine 25mg | Modafinil 400mg + Cocaine 25mg | Modafinil 0mg + Cocaine 50mg | Modafinil 200mg + Cocaine 50mg | Modafinil 400mg + Cocaine 50mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 2 (0.5) | 2 (0.5) | 2 (0.5) | 30 (5) | 28 (4) | 29 (3) | 44 (4) | 35 (4) | 35 (2) | 60 (3) | 55 (4) | 55 (4)

3. Secondary Outcome: Heart Rate
Description: Values for heart rate as a function of cocaine dose and modafinil maintenance condition.
Time Frame: 48 days
Population: Eight patients participated in each condition in a within-subjects fashion.
Measure: Mean (Standard Error); unit: BPM
Arm/Group | Modafinil 0mg + Cocaine 0mg | Modafinil 200mg + Cocaine 0mg | Modafinil 400mg + Cocaine 0mg | Modafinil 0mg + Cocaine 12mg | Modafinil 200mg + Cocaine 12mg | Modafinil 400mg + Cocaine 12mg | Modafinil 0mg + Cocaine 25mg | Modafinil 200mg + Cocaine 25mg | Modafinil 400mg + Cocaine 25mg | Modafinil 0mg + Cocaine 50mg | Modafinil 200mg + Cocaine 50mg | Modafinil 400mg + Cocaine 50mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
BPM | 88 (2) | 86 (2) | 91 (2) | 102 (3) | 101 (2.5) | 97 (3) | 130.5 (2) | 110 (3) | 115 (2.5) | 141 (2) | 125 (4) | 122 (2)

ADVERSE EVENTS:
Time Frame: 48 days
Groups:
- Modafinil 0 mg + Cocaine (0, 12, 25, and 50mg): During this within-subjects, alternating in-patient/outpatient 48-day study, participants were maintained on modafinil (0 mg/day) and a dose response of four doses of smoked cocaine (0, 12, 25, and 50mg).
- Modafinil 200 mg + Cocaine (0, 12, 25, and 50mg): During this within-subjects, alternating in-patient/outpatient 48-day study, participants were maintained on modafinil (200 mg/day) and a dose response of four doses of smoked cocaine (0, 12, 25, and 50mg).
- Modafinil 400 mg + Cocaine (0, 12, 25, and 50mg): During this within-subjects, alternating in-patient/outpatient 48-day study, participants were maintained on modafinil (400 mg/day) and a dose response of four doses of smoked cocaine (0, 12, 25, and 50mg).
Arm/Group | Modafinil 0 mg + Cocaine (0, 12, 25, and 50mg) | Modafinil 200 mg + Cocaine (0, 12, 25, and 50mg) | Modafinil 400 mg + Cocaine (0, 12, 25, and 50mg)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
This study is limited by the small, non-diverse sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes